CLINICAL TRIAL: NCT06308653
Title: A Phase 3, Randomized, Double-Blind, Multicenter Study to Evaluate the Efficacy, Safety, and Tolerability of Psilocybin in Adults With Major Depressive Disorder (MDD)
Brief Title: Psilocybin for Major Depressive Disorder (MDD)
Acronym: uAspire
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Usona Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PSIL301
Record Dates: First submitted 2024-03-06; First posted 2024-03-13 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Depressive Disorder, Major
Keywords: Psilocybin; Psychedelic; Depression; Major Depressive Disorder; MDD; Psychosocial; Psychoeducation; Set and Setting
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Psilocybin; microcrystalline cellulose; Psychiatric Rehabilitation

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive Psilocybin 25 mg, Psilocybin 5 mg, or inactive placebo under double-blind conditions. After the initial 6-week Double-blind Period, all participants will proceed into a 1-year Follow-up Period. During this 1-year Follow-up Period, eligible participants who meet pre-determined criteria may be offered open-label Psilocybin 25 mg in the context of a "Set and Setting" (SaS) Protocol.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The following roles will be blinded to the treatment group assignment in the Double-blind Period during the trial: Participant, Investigator, Site Personnel, Facilitators, Efficacy Raters (including Site Raters, Participant Raters, and Central Raters), Contract Research Organization (CRO) Staff, and Sponsor.
  All roles other than the Sponsor, CRO, and Ethics Committees will also be blinded to the randomization ratio and Patient Health Questionnaire-9 (PHQ-9) score for re-administration eligibility.
  The Central MADRS Rater will also be blinded to all aspects of the protocol and trial visit for each participant.
  Blinded trial site personnel will complete administration of the IP.
  Full blinding of trial personnel, Sponsor, and participants will be maintained until database lock at the conclusion of the trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Psilocybin 25 mg (Experimental): During the Double-blind Period, participants randomized to receive Psilocybin 25 mg will receive a single dose administered orally as a capsule and taken with water, along with the "Set and Setting" (SaS) Protocol.
  The "Set and Setting" (SaS) Protocol includes preparatory meetings with two Facilitators prior to dosing, a 7-10 hour dosing session in a comfortable room under the supervision of the same two Facilitators, and 4 hours of post-dose integration sessions with Facilitators. During the dosing session, participants are encouraged to wear eyeshades and listen to a curated playlist on headphones.
  Interventions: Drug: Psilocybin 25 mg
- Psilocybin 5 mg (Active Comparator): During the Double-blind Period, participants randomized to receive Psilocybin 5 mg will receive a single dose administered orally as a capsule and taken with water, along with the "Set and Setting" (SaS) Protocol.
  The "Set and Setting" (SaS) Protocol includes preparatory meetings with two Facilitators prior to dosing, a 7-10 hour dosing session in a comfortable room under the supervision of the same two Facilitators, and 4 hours of post-dose integration sessions with Facilitators. During the dosing session, participants are encouraged to wear eyeshades and listen to a curated playlist on headphones.
  Interventions: Drug: Psilocybin 5 mg
- Inactive Placebo (Placebo Comparator): During the Double-blind Period, participants randomized to receive inactive placebo will receive a single dose of Microcrystalline Cellulose (MCC) 25 mg administered orally as a capsule and taken with water, along with the "Set and Setting" (SaS) Protocol.
  The "Set and Setting" (SaS) Protocol includes preparatory meetings with two Facilitators prior to dosing, a 7-10 hour dosing session in a comfortable room under the supervision of the same two Facilitators, and 4 hours of post-dose integration sessions with Facilitators. During the dosing session, participants are encouraged to wear eyeshades and listen to a curated playlist on headphones.
  Interventions: Drug: Inactive Placebo
- Long-Term Follow-Up (Other): After the initial 6-week Double-blind Period, all participants will proceed to a 1-year Follow-up Period. Participants will be followed via in-clinic visits and telephone visits during which clinic staff will assess changes in MDD symptom severity and safety measures including concomitant medications, adverse events (AEs), and suicidal ideation and behavior.
  Participants will also engage in group psychosocial support sessions, including psychoeducation, throughout this period.
  Participants may also be eligible to receive open-label re-administration(s) of Psilocybin 25 mg under the "Set and Setting" (SaS) Protocol if re-administration eligibility criteria are met.
  Interventions: Drug: Psilocybin 25 mg; Behavioral: Psychosocial Support

INTERVENTIONS:
Drug: Psilocybin 25 mg — The Psilocybin used in this study is synthetically manufactured in a laboratory and meets quality specifications suitable for human research use. The active drug is encapsulated within a hydroxypropyl methylcellulose (HPMC) capsule and contains 25 mg of Psilocybin.
  Other Names: Psilocybine, Psilocibin, Indocybin
  Arms: Long-Term Follow-Up; Psilocybin 25 mg
Drug: Inactive Placebo — The inactive placebo is encapsulated within a hydroxypropyl methylcellulose (HPMC) capsule and contains 25 mg of Microcrystalline Cellulose (MCC). The MCC is synthetically manufactured in a laboratory and meets quality specifications suitable for human research use.
  Other Names: Microcrystalline Cellulose (MCC), Placebo
  Arms: Inactive Placebo
Drug: Psilocybin 5 mg — The Psilocybin used in this study is synthetically manufactured in a laboratory and meets quality specifications suitable for human research use. The active comparator is encapsulated within a hydroxypropyl methylcellulose (HPMC) capsule and contains 5 mg of Psilocybin.
  Other Names: Psilocybine, Psilocibin, Indocybin, Active Comparator
  Arms: Psilocybin 5 mg
Behavioral: Psychosocial Support — Psychosocial Support, including psychoeducation, begins after the Double-blind Period and continues throughout the 1-year Follow-up Period in order to enhance participant safety and maximize retention for the entire trial duration.
  Arms: Long-Term Follow-Up

SUMMARY:
Approximately 240 eligible adult participants (≥18 years old) who meet Diagnostic and Statistical Manual of Mental Disorders (DSM-5-TR) criteria for Major Depressive Disorder (MDD) will be enrolled. Participants will be randomly assigned to receive a single oral dose of Psilocybin 25 mg, Psilocybin 5 mg, or inactive placebo.

The purpose of this study is to evaluate the efficacy, safety, and tolerability of Psilocybin 25 mg versus placebo in adults with MDD, as assessed by the difference between groups in change in depressive symptoms from Baseline to Day 43 post-dose, and to characterize the durability of initial treatment effect and subsequent response to optional Psilocybin 25 mg re-administration(s) during the 1-year Follow-up Period.

DETAILED DESCRIPTION:
Double-blind Period:

Participants who show stable depression symptoms between Screening and Trial Baseline will be randomly assigned to receive a single oral dose of Psilocybin 25 mg, Psilocybin 5 mg, or inactive placebo.

Investigational Product (IP) will be administered in the context of a "Set and Setting" (SaS) Protocol for psychosocial support, comprised of 1) a period of preparation with Facilitators prior to dosing; 2) administration of IP in an aesthetically pleasing room under the supervision of two Facilitators; and 3) post-dose integration sessions during which participants will discuss their dosing experience with the Facilitators.

Trial outcome measures will assess depressive symptoms, functional disability, health-related quality of life, and clinical global impression of disease severity.

Long-term Follow-up Period:

After the initial 6-week Double-blind Period and completion of the post-dosing Trial Day 43 assessments, all participants will proceed into a 1-year Follow-up Period.

During the 1-year Follow-up Period, participants will be followed regularly by clinic staff to assess MDD symptom severity, functional disability, and health-related quality of life; long-term safety data will also be collected. In addition to scheduled clinic visits, clinic staff will contact participants by telephone every two weeks to assess for changes in MDD symptom severity, concomitant medications, adverse events (AEs), and suicidal ideation and behavior.

Participants who meet the pre-defined MDD severity criteria and meet all re-administration eligibility criteria may be offered re-administration(s) of open-label Psilocybin 25 mg administered under a "Set and Setting" (SaS) Protocol. Psychosocial support, including psychoeducation, is also incorporated in the long-term Follow-up Period.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years old.
* Able to swallow capsules.
* If of childbearing potential, agree to practice an effective means of birth control throughout the duration of the study.
* Meet the DSM-5-TR criteria for a diagnosis of major depressive disorder and are currently experiencing a major depressive episode of at least a 60-day duration at the time of Screening.
* Have at least moderate severity of depression symptoms at Screening and Trial Baseline.

Exclusion Criteria:

* Participants who are pregnant, who intend to become pregnant during the trial, or who are currently nursing.
* Have any of the following cardiovascular conditions: coronary artery disease, congenital long QT syndrome, cardiac hypertrophy, cardiac ischemia, congestive heart failure, clinically-relevant valvular heart disease, pulmonary hypertension, myocardial infarction, a clinically significant ECG abnormality, or tachycardia.
* Have elevated blood pressure.
* Have neurological conditions such as stroke, including transient ischemic attack, epilepsy, neurodegenerative disease (e.g., dementia, Parkinson's disease, Huntington's disease, amyotrophic lateral sclerosis, etc.), or brain tumor.
* Have severe hepatic or renal impairment.
* Have uncontrolled diabetes mellitus or unstable existing thyroid disorder.
* Are hepatitis or HIV positive.
* Have a positive urine drug test for illicit, non-prescribed, or prohibited substances.
* Meet DSM-5-TR criteria for schizophrenia spectrum or other psychotic disorders, including major depressive disorder with psychotic features ,bipolar disorder (types 1 or 2), antisocial personality disorder, borderline personality disorder or moderate or severe alcohol or drug use disorder
* Meet DSM-5-TR criteria for active post-traumatic stress disorder within 6 months prior to Screening.
* Have a first-degree relative with schizophrenia spectrum or other psychotic disorders, or bipolar I disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-03-13 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in central rater Montgomery-Asberg Depression Rating Scale (MADRS) total score from Baseline to Trial Day 43 | From Trial Baseline to Trial Day 43
  The MADRS is a clinician-rated scale designed to measure depression severity and to detect changes due to antidepressant treatment. The scale consists of 10 items, each of which is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), for a total possible score of 60. Higher scores represent a more severe condition. The total (composite) MADRS score is used as the endpoint.

SECONDARY OUTCOMES:
Change in central rater Clinical Global Impression-Severity (CGI-S) total score from Baseline to Trial Day 43 | From Trial Baseline to Trial Day 43
  The CGI-S is a 7-point scale, with a minimum score of 1 and a maximum score of 7, with higher scores representing more severe illness, that assesses the global severity of the participant's illness at the time of assessment relative to the clinician's past experience with patients who have the same diagnosis.
Change in on-site rater administered Sheehan Disability Scale (SDS) score from Baseline to post-dose Day 43 | From Trial Baseline to Trial Day 43
  The SDS is a composite of three self-rated items designed to measure the extent to which three major sectors in the patient's life are impaired by psychiatric symptoms, including depression. The SDS total score ranges from 0 to 30 with higher representing greater functional disability.

CONTACTS AND LOCATIONS:
Locations (29):
- United States (29):
  - University of Alabama Clinical Research Unit, Birmingham, Alabama
  - Preferred Research Partners-NWA, LLC, Fayetteville, Arkansas
  - Preferred Research Partners, Inc., Little Rock, Arkansas
  - Kadima Neuropsychiatry Institute, La Jolla, California
  - West LA VA Medical Center - Mental Health Department, Los Angeles, California
  - Pacific Neuroscience Institute (PNI) at Saint John's Physician Partners, Santa Monica, California
  - Psychedelic Science Institute, Santa Monica, California
  - Mountain View Clinical Research, Denver, Colorado
  - Connecticut Mental Health Center, Yale University, New Haven, Connecticut
  - Clinical Neuroscience Solutions Inc., Jacksonville, Florida
  - Innovative Clinical Research, Inc., Lauderhill, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Emory University, Atlanta, Georgia
  - CenExel iResearch, LLC, Decatur, Georgia
  - Great Lakes Clinical Trials, Chicago, Illinois
  - Johns Hopkins School of Medicine, Center for Psychedelic and Consciousness Research, Baltimore, Maryland
  - Sunstone Medical PC, Rockville, Maryland
  - Washington University School of Medicine, St Louis, Missouri
  - VA Nebraska Western Iowa Health Care System, Omaha, Nebraska
  - Global Medical Institutes, LLC; Princeton Medical Institute, Princeton, New Jersey
  - University of New Mexico (UNM) Interdisciplinary Substance Use and Brain Injury (ISUBI) Center, Albuquerque, New Mexico
  - NYU Clinical & Translational Science Institute, New York, New York
  - Bronx Veterans Research Foundation at the James J. Peters VAMC, The Bronx, New York
  - AIM Trials, LLC, Plano, Texas
  - Clinical Trials of Texas, LLC, San Antonio, Texas
  - Cedar Clinical Research, Draper, Utah
  - Cedar Clinical Research, Inc., Murray, Utah
  - Seattle Neuropsychiatric Treatment Center, Bellevue, Washington
  - VA Portland Health Care System, Vancouver, Washington

REFERENCES:
- [Result] Raison CL, Sanacora G, Woolley J, Heinzerling K, Dunlop BW, Brown RT, Kakar R, Hassman M, Trivedi RP, Robison R, Gukasyan N, Nayak SM, Hu X, O'Donnell KC, Kelmendi B, Sloshower J, Penn AD, Bradley E, Kelly DF, Mletzko T, Nicholas CR, Hutson PR, Tarpley G, Utzinger M, Lenoch K, Warchol K, Gapasin T, Davis MC, Nelson-Douthit C, Wilson S, Brown C, Linton W, Ross S, Griffiths RR. Single-Dose Psilocybin Treatment for Major Depressive Disorder: A Randomized Clinical Trial. JAMA. 2023 Sep 5;330(9):843-853. doi: 10.1001/jama.2023.14530. PMID 37651119
- [Derived] Palitsky R, Maples-Keller JL, Peacock C, Dunlop BW, Mletzko T, Grant GH, Raison CL, Chao S, Shub I, Mendelbaum-Kweller M, Smolyar L, Kaplan DM, Rothbaum BO, Zarrabi AJ. A critical evaluation of psilocybin-assisted therapy protocol components from clinical trial patients, facilitators, and caregivers. Psychotherapy (Chic). 2025 Sep;62(3):348-362. doi: 10.1037/pst0000551. Epub 2025 Jan 13. PMID 39804360